CLINICAL TRIAL: NCT07337278
Title: Effect of Lumbopelvic Rehabilitation Using Posturography Combined With Pelvic Floor Training on Urinary Incontinence in Women
Brief Title: Posturography Rehabilitation and Pelvic Floor Training on Urinary Incontinence in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed V University in Rabat (Other)
Responsible Party: Principal Investigator, Khaoula Mestour, Resident in Physical and Rehabilitation Medicine, Mohammed V University in Rabat
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UM5-MPR-2025-01
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence, Pelvic floor, Lumbopelvic static, Posturography
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two parallel groups: a combined pelvic floor muscle training and lumbopelvic postural rehabilitation group, and a pelvic floor muscle training alone group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Pelvic Floor Muscle Training and Posturography Rehabilitation (Experimental): Participants receive pelvic floor muscle training combined with lumbopelvic rehabilitation using posturography for a total duration of 12 weeks.
  Interventions: Behavioral: Pelvic Floor Muscle Training; Behavioral: Posturography Rehabilitation
- Pelvic Floor Muscle Training Alone (Active Comparator): Participants receive pelvic floor muscle training alone for a total duration of 12 weeks.
  Interventions: Behavioral: Pelvic Floor Muscle Training

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training — Pelvic floor training consists of voluntary contractions of the pelvic floor muscles, using short, rapid contractions combined with slow, sustained contractions, aimed at improving strength and endurance. Training is performed in supine and seated positions, with one supervised session per week at the hospital and three home sessions per week, over a total duration of 12 weeks.
Behavioral: Posturography Rehabilitation — Postural rehabilitation consists of seated exercises focusing on stability and mobility of the lumbopelvic region, using posturography. Sessions last 30 minutes, conducted twice weekly, over a total duration of 12 weeks.
  Arms: Combined Pelvic Floor Muscle Training and Posturography Rehabilitation

SUMMARY:
The goal of this clinical trial is to evaluate whether lumbopelvic postural rehabilitation combined with pelvic floor muscle training (PFMT) is more effective than PFMT alone in women with urinary incontinence. The main questions it aims to answer are:

* Does the addition of lumbopelvic postural rehabilitation improve the severity of urinary incontinence as measured by the ICIQ-UI-SF questionnaire?
* Does it improve urinary symptom profile, pelvic floor muscle strength, patient-reported overall improvement, and quality of life compared to PFMT alone?

Participants will be randomly assigned to one of two groups:

* Experimental group (Group A): PFMT (3 sessions/week) plus lumbopelvic postural rehabilitation (2 sessions/week) for 12 weeks.
* Control group (Group B): PFMT alone (3 sessions/week) for 12 weeks. Participants will perform pelvic floor exercises in supine and seated positions, with supervised sessions at the hospital and home exercises. Postural rehabilitation includes stability and mobility exercises for the lumbopelvic region using Posturography. Outcomes will be assessed at baseline, at 6 weeks, and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 65 years
* Presence of clinical signs of urinary incontinence (stress urinary incontinence and/or urge urinary incontinence and/or mixed urinary incontinence) diagnosed according to the International Continence Society (ICS) terminology
* USP (urinary symptom profile) scores for stress urinary incontinence and/or overactive bladder ≥ 1
* Normal neuro-perineal examination
* Written informed consent provided prior to participation in the study

Exclusion Criteria:

* Known detrusor overactivity or reduced bladder compliance of neurological origin
* Associated voiding dysfunction, defined as a Urinary Symptom Profile (USP) dysuria subscale score ≥ 1
* Known organic or morphological pathology of the lower urinary tract
* Pelvic organ prolapse grade II or higher according to the Pelvic Organ Prolapse Quantification system (POP-Q)
* Current urinary tract infection or vaginal infection
* Cognitive or visual impairments that may interfere with understanding or performing the exercise program
* Pregnant women or women within 10 months postpartum
* Anticholinergic medication use or hormone replacement therapy within the last 6 months
* Recent pelvic or abdominal surgery within the last 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) | 6 weeks and 12 weeks from start of intervention
  The primary outcome is the severity of urinary incontinence measured by the ICIQ-UI-SF. This validated questionnaire assesses frequency, quantity, and impact of leaks on quality of life. The overall score is obtained by adding up the 3 questions, ranging from 0 to 21, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | 6 weeks and 12 weeks from start of intervention
  PGI-I is a patient-reported questionnaire assessing overall improvement in urinary symptoms compared to baseline. Scores range from "considerably improved" to "considerably worsened".
Urinary Symptom Profile (USP) scores | 6 weeks and 12 weeks from start of intervention
  questionnaire enabling qualitative and quantitative analysis of urinary symptoms of stress urinary incontinence, overactive bladder, and dysuria. We used the subscores for stress urinary incontinence and overactive bladder.
Pelvic Floor Muscle Strength (Modified Oxford Scale) | 6 weeks and 12 weeks from start of intervention
  The modified Oxford scale assesses pelvic floor muscle strength through vaginal palpation and visual observation during maximum voluntary contraction. The classification ranges from 0 (no contraction) to 5 (strong contraction)
Incontinence Impact Questionnaire - Short Form (IIQ-7) | 6 weeks and 12 weeks from start of intervention
  IIQ-7 measures the impact of urinary incontinence on daily activities, social relationships, mobility, and emotional health. Each item is scored from 0 (not at all) to 3 (greatly), with higher total scores indicating greater impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ayachi Hospital, CHU Ibn Sina, Rabat, Rabat-Salé-Kénitra, Morocco

IPD SHARING:
Plan to Share IPD: No